CLINICAL TRIAL: NCT07403539
Title: Relationship Between Speech Perceptual Learning and Speech Production in Parkinson's Disease
Brief Title: Speech Learning and Speech Production in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Mishaela DiNino, Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00008661
Record Dates: First submitted 2026-01-27; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Parkinson's Disease
Keywords: speech perception; communication; learning
MeSH Terms: conditions — Parkinson Disease; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Learning and Discrimination (Experimental): Behavioral interventions will be administered, including speech intensity learning, speech intensity discrimination, speech rate learning, and speech rate discrimination
  Interventions: Behavioral: Intensity learning; Behavioral: Intensity discrimination; Behavioral: Rate learning; Behavioral: Rate discrimination

INTERVENTIONS:
Behavioral: Intensity learning — Participants will be asked to pair sentences that vary in their sound intensity to one of three colored squares (red, yellow, or blue)
Behavioral: Intensity discrimination — Participants will hear two sentences that are either the same or different in their sound intensity and will be asked to indicate whether the sentences were of the same or different intensities
Behavioral: Rate learning — Participants will be asked to pair sentences that vary in their spoken rate to one of three colored squares (red, yellow, or blue)
Behavioral: Rate discrimination — Participants will hear two sentences that are either the same or different in their spoken rate and will be asked to indicate whether the sentences were of the same or different rates

SUMMARY:
Parkinson's disease, a common movement disorder that results from a breakdown in the brain, often leads to challenges with talking, but less is known about the relationship between difficulties with talking and difficulties with learning to understand speech. By linking these two abilities in individuals with Parkinson's disease using a precision medicine approach, this project seeks to build a basis for new therapies that help people with Parkinson's disease both understand better and speak more clearly.

DETAILED DESCRIPTION:
In the context of speech-language therapy, Parkinson's disease (PD) is typically associated with its consequences on speech production. Interventions generally focus on learning or relearning skills to accomplish successful production. However, the disease itself, as well as patient responses to interventions, are variable. Individuals differ widely in how typical their speech output is before intervention and in how much they learn from treatment. One plausible explanation for this variation comes from a less-studied aspect of speech and language in PD: speech perception, especially speech perceptual learning. There is a key gap in the PD literature about whether people who produce atypical rate and intensity properties in their own speech also find it more difficult to learn rate and intensity properties from others' speech. There is, therefore, a critical need for a full understanding of the relationship between speech production and speech perceptual learning in PD. The long- term goal of this research program is to systematically interrogate the relationship between speech learning and production in people with PD and to leverage that knowledge to promote effective communication. The overall objective of this project is to use acoustic measures to determine how challenges with speech perception or learning can predict individual differences in speech production. The central hypothesis is that individual differences between people with PD in speech perception or learning can predict individual differences between people with PD in speech production. This project adopts an individual differences approach to investigate two major aims: (1) relating individual differences in the perceptual learning of speech rate to the production of speech rate, and (2) relating individual differences in the perceptual learning of intensity to the production of intensity. To investigate these aims, each participant will record a speech sample and conduct tasks that involve learning regularities in rate or intensity in the speech of others. Participants will also complete tasks that require the ability to distinguish between sentences based on their rate and intensity. Participants' speech samples will additionally be judged by naive listeners to assess the samples' intelligibility and the effort that it takes to understand the speakers. If individual differences in perceptual learning predict individual differences in production, then differences in speech perception may predict differences in speech-language therapy outcomes that could be targeted to patient needs. A precision medicine approach would allow for interventions that titrate the amount, level, and type of intervention on an individualized basis to make sure that treatments are focused on participants who will respond to them in dosages that they will benefit from. For instance, a therapist could provide speech perception training to accelerate outcomes of production-related treatments. Furthermore, by applying more naturalistic measures of speech perception to this population, especially ones that rely on participants to change over the course of a session, this project provides an innovative opportunity to examine the sensory and perceptual consequences of PD and to link those to better-documented motor outcomes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Native speaker of North American English
* Use a drug that includes levodopa
* Resident of the United States

Exclusion Criteria:

* Any history of language, hearing or speech disorder outside of Parkinson's disease
* Other gross neurological impairment such as Alzheimer's disease or stroke
* Significant hearing loss and/or use of a hearing aid or cochlear implant

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean dB SPL | Day 1
  The mean speech intensity (in dB SPL) will be assessed using a recording of spoken sentences and a spoken paragraph.
Standard deviation dB SPL | Day 1
  The standard deviation of participant's speech intensity (in dB SPL) will be assessed using a recording of spoken sentences and a spoken paragraph.
Speaking rate | Day 1
  The speaking rate (in syllables/second) will be assessed using a recording of spoken sentences and a spoken paragraph.
Articulation rate | Day 1
  The articulation rate (in syllables/second after removing pauses) will be assessed using a recording of spoken sentences and a spoken paragraph.
Unfilled pause time | Day 1
  The unfilled pause time (in seconds of pause) will be assessed using a recording of spoken sentences and a spoken paragraph.

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified speech perception and speech production data from individual participants
Supporting Information: Study Protocol, SAP
Time Frame: Information will be available at the conclusion of data collection and will be available indefinitely
Access Criteria: Data and supporting material will be available on the Open Science Framework, a database that is open to the general public